CLINICAL TRIAL: NCT01300442
Title: Fundamentation of TEDS Protocol in Healthy Subjects and Its Application in COPD Patients
Brief Title: Effects of Transcutaneous Electrical Diaphragmatic Stimulation on Respiratory Variables in COPD Patients
Acronym: COPD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Dr. Dirceu Costa, PNPD / CNPq
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DC1901-PNPD
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-01

CONDITIONS: COPD
Keywords: chronic obstructive pulmonary disease; diaphragm; electrical stimulation; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Experimental): The transcutaneous electrical diaphragmatic stimulation will be applied in healthy and COPD subjects.
  Interventions: Other: TEDS in healthy patients
- Chronic Obstructive Pulmonary Disease (Experimental): The intervention will be the TEDS in patients with Chronic Obstructive Pulmonary Disease (COPD)
  Interventions: Other: TEDS in COPD patients

INTERVENTIONS:
Other: TEDS in COPD patients — For the TEDS (transcutaneous electrical diaphragmatic stimulation) the electrical current is pulsed, biphasic and symmetric, with the following parameters: frequency of 30 Hertz; 0.4ms phase width, rise time of 0.7 seconds; respiratory rate of 14 rpm; intensity is the minimum necessary to obtain diaphragm muscle contraction. Four silicone-carbon electrodes (3x5cm) were placed on the skin with gel and micropore tape. Two electrodes were located on each side of the thorax, specifically in the 3rd intercostal space near the xyphoid region and in the 7th intercostal space, on the mid-axillary line. Each session had duration of approximately 30 minutes and the subjects were instructed to co-ordinate breathing with the pulsing of the electrical current.
  Other Names: The equipment is the Dualpex 961 model Phrenics (Quark®).
  Arms: Chronic Obstructive Pulmonary Disease
Other: TEDS in healthy patients — For the TEDS (transcutaneous electrical diaphragmatic stimulation) the electrical current is pulsed, biphasic and symmetric, with the following parameters: frequency of 30 Hertz; 0.4ms phase width, rise time of 0.7 seconds; respiratory rate of 14 rpm; intensity is the minimum necessary to obtain diaphragm muscle contraction. Four silicone-carbon electrodes (3x5cm) were placed on the skin with gel and micropore tape. Two electrodes were located on each side of the thorax, specifically in the 3rd intercostal space near the xyphoid region and in the 7th intercostal space, on the mid-axillary line. Each session had duration of approximately 30 minutes and the subjects were instructed to co-ordinate breathing with the pulsing of the electrical current.
  Other Names: The equipment is the Dualpex 961 model Phrenics (Quark®).
  Arms: Control

SUMMARY:
Transcutaneous electrical diaphragmatic stimulation (TEDS) has been used to improve respiratory muscle strength in patients with respiratory muscles weakness. However, this physiotherapeutic resource has not been studied in chronic obstructive pulmonary disease (COPD) yet. The objective of this study is to evaluate the respiratory pattern during the session of TEDS besides its effect in respiratory muscle strength and in spirometric variables as much healthy patients as in COPD patients. Methods: healthy and COPD patients are selected and submitted to TEDS treatment. The plethysmographic analysis (LifeShirt System - VivoMetric), respiratory muscle strength and spirometry will be made. The hypothesis is that the TEDS can helps COPD patients that shows respiratory muscle weakness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable COPD (diagnosed by accepted criteria)
* Healthy patients

Exclusion Criteria:

* FOR THE COPD PATIENTS:
* Over 80 years of age
* History of recent exacerbation
* Patients with pacemakers
* Uncontrolled arterial hypertension
* Requiring home oxygen therapy.
* FOR THE HEALTHY PATIENTS:
* Pulmonary diseases
* Cardiovascular diseases
* Orthopedic diseases
* Neurologic diseases.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-04 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength and spirometry | 06 weeks
  Respiratory muscle strength: maximal inspiratory pressure (cH2O) and maximal expiratory pressure (cH2O) by manovacuometer (Gerar®) Spirometry by Spirometer EasyOne®

SECONDARY OUTCOMES:
Respiratory pattern | During the session of transcutaneous electrical diaphragmatic stimulation
  Inductance pletismography by LifeShirt® (VivoMetrics). The variables are: inspiratory tidal volume (ViVol); expiratory tidal volume (VeVol); minute ventilation (VE) in liters; inspiratory time (Ti); expiratory time (Te); total breath time (Tt) in seconds; phase relation during inspiration (PhRIB); phase relation during expiration (PhREB); phase relation of the entire breath (PhRTB) and phase angle (PhAng) in percentage (%).

CONTACTS AND LOCATIONS:
Overall Officials: Dirceu Costa, PhD, Study Director — UFSCar
Locations (1):
- UFSCar, São Carlos, São Paulo, Brazil

REFERENCES:
- [Derived] Cancelliero-Gaiad KM, Ike D, Pantoni CB, Mendes RG, Borghi-Silva A, Costa D. Acute effects of transcutaneous electrical diaphragmatic stimulation on respiratory pattern in COPD patients: cross-sectional and comparative clinical trial. Braz J Phys Ther. 2013 Nov-Dec;17(6):547-55. doi: 10.1590/S1413-35552012005000121. Epub 2013 Nov 14. PMID 24271095